CLINICAL TRIAL: NCT02231528
Title: Interest of Ultrasound Coupled to a Guidance System (GPS) for Central Venous Catheters (CVC) Insertion.
Acronym: VVC and GPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1230
Record Dates: First submitted 2014-08-27; First posted 2014-09-04 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Surgery
Keywords: anesthesia; central venous catheter; jugular vein; ultrasound guidance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Use of ultrasound with active GPS (Experimental)
  Interventions: Device: Use of ultrasound with active GPS
- Use of ultrasound with inactive GPS (Active Comparator)
  Interventions: Device: Use of ultrasound with inactive GPS

INTERVENTIONS:
Device: Use of ultrasound with active GPS — CVC insertion with ultrasound with active GPS function and appropriate needles
  Arms: Use of ultrasound with active GPS
Device: Use of ultrasound with inactive GPS — CVC insertion with ultrasound with inactive GPS function and conventional needles
  Arms: Use of ultrasound with inactive GPS

SUMMARY:
The GPS system would simplify the technical implementation of central venous catheter under ultrasound guidance. We can assume that the introduction of deep venous pathways (as a reference, the internal jugular) will be faster, and this, whatever the level of expertise. By checking this hypothesis, this technique could be applied to much less frequent situations establishment of difficult central venous catheters (hemodynamic status precarious, hypovolemia, or cardiac arrest).

The main objective of this study is to evaluate the time savings provided by the ultrasound assisted GPS guidance for installing central venous catheters in the internal jugular. Central venous catheters are inserted in the operating room under conditions scheduled in advance that is to say outside emergency. The installation time for the central venous catheter is compared with that obtained by using the ultrasound machine without the GPS guide ("conventional" technique).

DETAILED DESCRIPTION:
The techniques of reference for the central venous access (internal jugular, subclavian or femoral) are based on anatomical landmarks and the low probability of anatomical variations. With these techniques, the central venous puncture, with Seldinger method, is associated to complications both in adults and in children (pneumothorax, hemothorax, infection, thrombosis, arterial puncture, inappropriate location). The frequency of these adverse events is highly variable and ranges between 1 and 20% of central venous catheters in place. Ultrasound, visualizing anatomical structures before (echo tracking) or during (ultrasound guidance) the puncture, improves about 80% the success of the first puncture, and decreases by 50% the complications. The ultrasound guidance is better than echo tracking to reduce the time of implementation of the central venous catheter. However, this technique requires more practice. On the other hand, visualization of the needle path is not always easy especially for the subclavian access, because it requires a puncture in the ultrasound plane.

GPS system (Guidance Positioning System) is an original system of guidance. This is a simple navigation system for projecting the theoretical position of the puncture needle in the ultrasound plane. The guidance system consists of a receiver and two motion sensors. The receiver is connected to the system. A motion sensor is incorporated into the end of the needle. Another motion sensor is located within the ultrasound probe. The relative positions and the axes of the needle and the ultrasound probe are transmitted with coordinates in three dimensions.

The puncture can be carried out of the plane (ultrasound probe perpendicular to the axis puncture) and the direct visualization of the needle is not necessary. Before the puncture, the end of the needle is placed on the skin. The direction and the axis of the needle relative to the skin are adjusted, before the puncture, depending on the position of the target to be achieved, displayed by a mark on the screen. Throughout the puncture, a projected image of the needle is displayed on the screen.

ELIGIBILITY:
Inclusion Criteria:

* Adults 2 sexes
* Age> 18years
* Indication for placing a central venous catheter in internal jugular
* Scheduled installation

Exclusion Criteria:

* Persons referred to in Articles L. 1121-5 to L. 1121-8 Code of Public Health,
* Lack of coverage by social security
* Refusal of patient consent
* Contraindication for placement of a central venous catheter in internal jugular
* Emergency
* Pregnancy
* Doppler data from the supra-aortic trunks if it exists (eg bilateral carotid stenosis)
* Pacemaker, defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Time required for CVC insertion | at the end of the insertion of the guide wire, an average of one and a half minutes after the beginning of the procedure

SECONDARY OUTCOMES:
Total number of puncture | at the end of the insertion of the guide wire, an average of one and a half minutes after the beginning of the procedure
Complication rate in the superior vena cava territory | At 24 hours
  Complication rate secondary to cannulation in the territory superior vena cava: arterial puncture, subcutaneous hematoma, pneumothorax, difficulty progression of the guide, aberrant pathway, transfixion of the vein
Insertion failure rate | at the end of the insertion of the guide wire, an average of one and a half minutes after the beginning of the procedure
  Failure is defined as the necessity to change anatomical site despite the visualization of the vein or stop using the GPS function

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ALBALADEJO, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU de Grenoble, Grenoble, France

REFERENCES:
- [Background] Graham AS, Ozment C, Tegtmeyer K, Lai S, Braner DA. Videos in clinical medicine. Central venous catheterization. N Engl J Med. 2007 May 24;356(21):e21. doi: 10.1056/NEJMvcm055053. No abstract available. PMID 17522396
- [Background] Hind D, Calvert N, McWilliams R, Davidson A, Paisley S, Beverley C, Thomas S. Ultrasonic locating devices for central venous cannulation: meta-analysis. BMJ. 2003 Aug 16;327(7411):361. doi: 10.1136/bmj.327.7411.361. PMID 12919984
- [Background] Randolph AG, Cook DJ, Gonzales CA, Pribble CG. Ultrasound guidance for placement of central venous catheters: a meta-analysis of the literature. Crit Care Med. 1996 Dec;24(12):2053-8. doi: 10.1097/00003246-199612000-00020. PMID 8968276
- [Background] Hosokawa K, Shime N, Kato Y, Hashimoto S. A randomized trial of ultrasound image-based skin surface marking versus real-time ultrasound-guided internal jugular vein catheterization in infants. Anesthesiology. 2007 Nov;107(5):720-4. doi: 10.1097/01.anes.0000287024.19704.96. PMID 18073546
- [Background] American Society of Anesthesiologists Task Force on Central Venous Access; Rupp SM, Apfelbaum JL, Blitt C, Caplan RA, Connis RT, Domino KB, Fleisher LA, Grant S, Mark JB, Morray JP, Nickinovich DG, Tung A. Practice guidelines for central venous access: a report by the American Society of Anesthesiologists Task Force on Central Venous Access. Anesthesiology. 2012 Mar;116(3):539-73. doi: 10.1097/ALN.0b013e31823c9569. No abstract available. PMID 22307320